CLINICAL TRIAL: NCT00723619
Title: Investigation of Lungfunction Normal Values in Children and Adolescent in Germany
Brief Title: Investigation of Lungfunction Normal Values in Children and Adolescent in Germany (Spirometry, Ultrasonic Pneumography and Exhaled NO)
Acronym: LUNOKID-Studie
Status: Completed | Type: Observational
Sponsor: Marien Hospital Wesel (Other)
Collaborators: Hannover Medical School (Other); Heinrich-Heine University, Duesseldorf (Other)
Responsible Party: Prof. Dr. D. Berdel, Marienhospital Wesel, Forschungsintitut zur Prävention von Allergien und Atemwegserkrankungen im Kindes- und Jugendalter
Other Study IDs: 2007067
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2010-02-17 (Estimated); Status verified 2008-07

CONDITIONS: Healthy
Keywords: asthma; spirometry; FENO; normal values for spirometry in childhood; normal values for FENO in childhood
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Children and adolescent from German schools in the region Wesel, Hannover and Düsseldorf, selected via special school lists

SUMMARY:
Synopsis: LUNOKID-Study

Investigation of Lung function Normal Values in Children and Adolescent in Germany

For the diagnostic work-up of childhood airway diseases lungfunction measurements play an important role. As childhood represents a period of continuous development and growth, not only is body size and weight increasing and body composition changing with age, but also is the lung developing both in size and airway differentiation. Results from lung function measurements in children and adolescents have thus to be related to lung function data which have been determined in a normal healthy age-matched childhood population. The quality of the reference values is therefore crucial for the interpretation of lung function results.

The reference values for children that are used today have been created between around the 1970th or 1980th, although the development and body size of children in the last decades has considerably changed and accelerated.

The aim of the LUNOKID study is to create new reference values for lung function measures in healthy children aged 4 to 18 years. Measurements will be performed in schools and "kindergartens" in 3 regions of Germany (Wesel, Düsseldorf, Hannover).

A modified ISAAC questionnaire will be distributed to the parents to get information on the family´s and child´s health history with regard to atopy, airway diseases or other diseases that could influence the lung function results. A clinical examination on the day of lung function performance should exclude acute infections or other diseases. Parents will have to give informed consent to the study.

Study personal, especially trained in the lung function unit of the University Hannover, is going to do all examination and lung function measures during the normal school hours at the sites of the schools and kindergartens.

The following measurements will be performed according to the respective SOPs:

* Body weight and hight
* Exhaled NO, using the NIOX -MINO in children from the age of 5 years onwards, in 4 years old children using the off-line method (both Aerocrine)
* Spirometry including Flow volume curves (Parameter FEV1, FEV0.5, FEV 0.75, PEF, FVC, MEF 25, MEF 50, MEF 75) using a Spirometer by the company ndd Medizintechnik AG, Zürich
* Ultrasonic pneumography (UPG) (tidal breathing), ndd Medizintechnik AG, Zürich

It is planned to have 50 valid measurements per gender and age group. Considering that about 50 % of the children (and 50-75% of the 4 years´old) have to be excluded for the "normal reference analysis" either for health reasons or because the lung function measurement cannot be correctly performed. The investigators therefore calculate to included in the study around 3300 children.

All data will be gathered and managed in a central database in the IUF in Düsseldorf. The statical analysis will include regression analyses to calculate the reference values.

It is planned to have the new reference values included in the guidelines for diagnostic and management of asthma in childhood, and in the software of lung function equipment. By now, the study is approved by the Ethical Committee responsible for the PI in Wesel.

DETAILED DESCRIPTION:
For detailed description please contact:

forschungsinstitut1@marien-hospital-wesel.de

ELIGIBILITY:
Inclusion Criteria:

* All children from a selected classes, which have an informed consent and an answered questionnaire

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: children and adolescents from classes and kindergarten in the regions Wesel,Düsseldorf and Hannover
Sampling Method: Probability Sample
Enrollment: 2007 (Actual)
Dates: Start 2007-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dietrich Berdel, Prof. Dr., Study Chair — Marien Hospital Wesel
Locations (1):
- Marien Hospital Wesel gGmbH, Wesel, North Rhine-Westphalia, Germany